CLINICAL TRIAL: NCT01905059
Title: Multicenter, International, Prospective, Phase III, Randomized, Superiority Trial Comparing Two Maintenance Strategies With Mono or Bi-therapy of Protease Inhibitors With or Without Lamivudine in Virologically Suppressed HIV Patients on Second Line Antiretroviral Treatment Over a Period of 96 Weeks in Africa (Dakar, Bobo Dioulasso, Yaounde)
Brief Title: Evaluation of a Maintenance Strategy With Protease Inhibitors With or Without Lamivudine in Virologically Suppressed HIV Patients on Second Line Antiretroviral Treatment in Africa
Acronym: MOBIDIP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 12286MOBIDIP
Record Dates: First submitted 2013-07-15; First posted 2013-07-23 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: HIV Infection
Keywords: HIV infection; second line ART; maintenance strategies; Protease inhibitors; mono or bi-therapy
MeSH Terms: conditions — HIV Infections | interventions — Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- monoPI - boosted lopinavir or boosted darunavir (Active Comparator): boosted lopinavir (LPV/rtv 200/50 mg 2 tbs BID) or boosted darunavir (DRV 400 mg 2 tbs plus RTV 100 mg QD)
  This arm has been stopped on advise of DSMB (approved by Scientific Committee), patients are switched to standard second line triple therapy and followed until the end of the study at week 96.
  Interventions: Drug: monoPI - boosted lopinavir or boosted darunavir
- bi therapy - (boosted lopinavir or darunavir) + lamivudine (Active Comparator): boosted lopinavir (LPV/rtv 200/50 mg 2 tbs BID) with lamivudine 300 mg QD or boosted darunavir (DRV 400 mg 2 tbs plus RTV 100 mg QD)with lamivudine 300 mg QD
  Interventions: Drug: bi therapy - (boosted lopinavir or boosted darunavir) + lamivudine

INTERVENTIONS:
Drug: monoPI - boosted lopinavir or boosted darunavir — boosted lopinavir (LPV/rtv 200/50 mg 2 tbs BID) or boosted darunavir (DRV 400 mg 2 tbs plus RTV 100 mg QD) This arm was stopped by the Scientific Committee on advise of the DSMB after interim analysis showing increased risk of failure for these participants. Participants are switched to standard second line triple therapy and will be followed until the last visit at week 96.
  Other Names: Protease Inhibitor monotherapy; boosted darunavir monotherapy; boosted lopinavir monotherapy
  Arms: monoPI - boosted lopinavir or boosted darunavir
Drug: bi therapy - (boosted lopinavir or boosted darunavir) + lamivudine — boosted lopinavir (LPV/rtv 200/50 mg 2 tbs BID) with lamivudine 300 mg QD or boosted darunavir (DRV 400 mg 2 tbs plus RTV 100 mg QD)with lamivudine 300 mg QD. This arm is going on, patients will be followed on this intervention until the end of the study at week 96
  Other Names: bi therapy; PI + 3TC; Boosted Protease Inhibitors plus lamivudine; LPV/r with lamivudine and DRV/r with lamivudine
  Arms: bi therapy - (boosted lopinavir or darunavir) + lamivudine

SUMMARY:
Multicenter, randomized, superiority trial to evaluate efficacy of a mono or bi-therapy of protease inhibitors with or without lamivudine over a period of 96 weeks. The primary outcome will be the failure rate at 96 weeks. This study will include 260 participants, former participants of the 2LADY trial. It will be carried out in Yaoundé, Bobo Dioulasso and Dakar.

DETAILED DESCRIPTION:
Justification: The interest of treating HIV infection with a single molecule has been clear for a long time. Many clinical trials have been testing the efficacy of such a strategy, mainly using a boosted protease inhibitor (PI). Despite the remaining doubts about low level viremia, viral control in reservoirs, durability of the effect, the trials showed attractive results with an absolute increase in the risk of virological failure between 2% and 13% compared to the standard of care and a possible decrease in costs and toxicity.

In resource-limited countries the interest of treatment simplification is even more important: decrease in costs, toxicity (often poorly monitored), number of pills taken per day, etc. In addition, for patients in second line for whom some kind of resistance to NRTI is highly probable, the interruption of the second line NRTI could help to avoid the accumulation of mutations in the RT in the presence of residual low level replication, sparing future treatment options.

The 184 mutation of the retro-transcriptase which causes resistance to lamivudine/emtricitabine seems to hinder viral replication. The persistence of this mutation could eventually facilitate the action of PI monotherapy while protecting patients from further mutations. The choice of viral load (VL) threshold for the diagnosis of failure in resource-limited countries is not easy, the 2LADY trial used in clinical practice, the threshold of 1000 copies/ml which allows genotyping for evidence of mutations. This value will probably be selected as a reference value by the WHO in its next recommendations. To minimize the risk of viral escape and the development of resistances in the MOBIDIP study the threshold of 200 copies/ml has been chosen for the switch to monotherapy and of 500 copies/ml for the definition of failure.

Principal objective: To evaluate the failure rate at 96 weeks of a PI monotherapy with or without lamivudine, in HIV positive patients on second line treatment (ART) for at least 48 weeks, and with a VL of less than 200 copies/ml in Africa (Yaoundé, Bobo Dioulasso, Dakar).

Specific objectives: To evaluate:

* viral efficacy at a threshold of 50 copies/ml at 48 and 96 weeks,
* failure rate at 500 copies/ml after 24 weeks from the reintroduction of NRTI backbone in case of monotherapy failure,
* clinical and immunological outcomes,
* development of mutations,
* tolerance and impact on metabolic profile and
* neuro-cognitive disorders,
* adherence

Methods: multicenter, randomized, superiority trial to evaluate efficacy of a mono or bi-therapy of protease inhibitors with or without lamivudine over a period of 96 weeks. The primary outcome will be the failure rate at 96 weeks. Failure is defined as: 1) viral load ≥500 copies/ml, 2) reintroduction of NRTI backbone, 3) interruption of the PI. A sample of 260 participants is planned.

Schedule: After approval by national Ethical committees and national authorities, patients followed in 2LADY trial for at least 48 weeks, and presenting the eligibility criteria, will stop their NRTI backbone and be randomized (over 6 months) to add or not lamivudine to their PI monotherapy. All patients will be followed for 96 weeks. In case of viral load above 500 copies/ml during the study, the original NRTI backbone will be re-introduced and the patient will be followed for an extra 24 weeks to verify viral response. The complete trial is due to last 3 years.

Expected results: This study will allow the validation of a maintenance strategy for patients in second line ART less expensive and toxic. In addition results could be used to guide clinical practice for physicians in resources poor countries

In march 2016 an interim analysis asked by the DSMB showed increased risk of failure in the monotherpay arm and the arm was stopped. Participant are switched on standard second line triple therapy and followed until Week 96. Participant on dual therapy continue their follow up. Comparative analysis are planned for data on week 60 visit (last visit with all participants on the randomized treatment).

ELIGIBILITY:
Inclusion Criteria:

* HIV infection on second line treatment in the 2lady trial for at least 48 weeks
* VL ≤ 200 copies/ml since at least 6 months
* No change in ART in the last 3 months previous to the study
* CD4> 100 cells/ml
* Signed informed consent
* Adherence >90

Exclusion Criteria:

* Previous viral failure (at least 2 consecutive HIV RNA >1000 copies/ml) while receiving a PI
* Ongoing pregnancy and breast feeding women
* HBsAg positive patients
* opportunistic infection or any severe or progressive disease ongoing or treated in the 3 months before screening
* Subject who in the investigator's opinion is unable to complete the study
* History or symptoms of HIV encephalopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2014-02; Primary Completion 2016-04 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in virological failure | 96 weeks
  Number of patients with a treatment failure. Definition of treatment failure: 1) viral load ≥ 500 copies/ml confirmed in 2 samples with 1 month interval, or 2) the reintroduction of the two NRTIs or 3) interruption of the boosted PI.

SECONDARY OUTCOMES:
Treatment failure after reintroduction of the baseline NRTI backbone regimen | 24 weeks from reintroduction NRTI regimen
  Number of patients in virological failure after reintroduction NRTI regimen. Treatment failure defined by viral load > 200 and/or > 500 copies/ml within 24 weeks from the reintroduction of the baseline NRTI backbone regimen
Virological response | 48 weeks
  Number of patient with VL < 50 copies/ml
The viral resistance | 24 weeks from reintroduction NRTI regimen
  The frequency of resistance mutations in the case of treatment failure
The clinical course of the HIV infection | Inclusion to 96 weeks
  Numbers of : AIDS events, non-AIDS events, death, adverse events
The Immune response | Between the inclusion and 96 weeks
  The variation in the level of circulating CD4+ lymphocytes
Tolerability | Between the inclusion and 96 weeks
  Changes to the parameters in baseline lipid profile, renal function and bone mineral density
Assessment of the adherence | 96 weeks but an average of mesures of each visits
  Adherence is considered high if consumption is greater than or equal to 95%, average if it is between 80 and 95% and low if it is less than 80%.
  It is measured at each visit, by means of a questionnaire and by tablet count.
Changes in anthropometric measures | between the inclusion and 96 weeks
  Changes to the following anthropometric measurements: waist circumference, hip circumference and thigh circumference
Assessment neurocognitive functions | 96 weeks
  screening questions (EACS Guidelines)
virological response | 96 weeks
  Number of patient with VL < 50 copies/ml

CONTACTS AND LOCATIONS:
Overall Officials: Koulla Shiro Sinata, Prof, Principal Investigator — University of Yaounde; Sawadogo Adrien, Dr, Principal Investigator — Hopital de Jour CHU Bobo Dioulasso; Ndour Cheik Tidiane, Prof, Principal Investigator — Service Maladies Infectieuses CHU Fann Dakar; Ciaffi Laura, Dr, Principal Investigator — UMI 233 IRD Montpellier
Locations (5):
- Day Care Center CHU Sanou Sauro, Bobo-Dioulasso, Burkina Faso
- Cameroon (2):
  - Central Hospital, Yaoundé
  - Military Hospital, Yaoundé
- Senegal (2):
  - CRCF Hopital de Fann, Dakar
  - CTA CHU de Fann, Dakar

REFERENCES:
- [Background] Arribas JR, Pulido F, Delgado R, Lorenzo A, Miralles P, Arranz A, Gonzalez-Garcia JJ, Cepeda C, Hervas R, Pano JR, Gaya F, Carcas A, Montes ML, Costa JR, Pena JM. Lopinavir/ritonavir as single-drug therapy for maintenance of HIV-1 viral suppression: 48-week results of a randomized, controlled, open-label, proof-of-concept pilot clinical trial (OK Study). J Acquir Immune Defic Syndr. 2005 Nov 1;40(3):280-7. doi: 10.1097/01.qai.0000180077.59159.f4. PMID 16249701
- [Background] Pulido F, Arribas JR, Delgado R, Cabrero E, Gonzalez-Garcia J, Perez-Elias MJ, Arranz A, Portilla J, Pasquau J, Iribarren JA, Rubio R, Norton M; OK04 Study Group. Lopinavir-ritonavir monotherapy versus lopinavir-ritonavir and two nucleosides for maintenance therapy of HIV. AIDS. 2008 Jan 11;22(2):F1-9. doi: 10.1097/QAD.0b013e3282f4243b. PMID 18097218
- [Background] Cameron DW, da Silva BA, Arribas JR, Myers RA, Bellos NC, Gilmore N, King MS, Bernstein BM, Brun SC, Hanna GJ. A 96-week comparison of lopinavir-ritonavir combination therapy followed by lopinavir-ritonavir monotherapy versus efavirenz combination therapy. J Infect Dis. 2008 Jul 15;198(2):234-40. doi: 10.1086/589622. PMID 18540803
- [Background] Cahn P, Montaner J, Junod P, Patterson P, Krolewiecki A, Andrade-Villanueva J, Cassetti I, Sierra-Madero J, Casiro AD, Bortolozzi R, Lupo SH, Longo N, Rampakakis E, Ackad N, Sampalis JS. Pilot, randomized study assessing safety, tolerability and efficacy of simplified LPV/r maintenance therapy in HIV patients on the 1 PI-based regimen. PLoS One. 2011;6(8):e23726. doi: 10.1371/journal.pone.0023726. Epub 2011 Aug 19. PMID 21886816
- [Background] Vernazza P, Daneel S, Schiffer V, Decosterd L, Fierz W, Klimkait T, Hoffmann M, Hirschel B. The role of compartment penetration in PI-monotherapy: the Atazanavir-Ritonavir Monomaintenance (ATARITMO) Trial. AIDS. 2007 Jun 19;21(10):1309-15. doi: 10.1097/QAD.0b013e32814e6b1c. PMID 17545707
- [Background] Gutmann C, Cusini A, Gunthard HF, Fux C, Hirschel B, Decosterd LA, Cavassini M, Yerly S, Vernazza PL; Swiss HIV Cohort Study (SHCS). Randomized controlled study demonstrating failure of LPV/r monotherapy in HIV: the role of compartment and CD4-nadir. AIDS. 2010 Sep 24;24(15):2347-54. doi: 10.1097/QAD.0b013e32833db9a1. PMID 20802298
- [Background] Katlama C, Valantin MA, Algarte-Genin M, Duvivier C, Lambert-Niclot S, Girard PM, Molina JM, Hoen B, Pakianather S, Peytavin G, Marcelin AG, Flandre P. Efficacy of darunavir/ritonavir maintenance monotherapy in patients with HIV-1 viral suppression: a randomized open-label, noninferiority trial, MONOI-ANRS 136. AIDS. 2010 Sep 24;24(15):2365-74. doi: 10.1097/QAD.0b013e32833dec20. PMID 20802297
- [Background] Arribas JR, Horban A, Gerstoft J, Fatkenheuer G, Nelson M, Clumeck N, Pulido F, Hill A, van Delft Y, Stark T, Moecklinghoff C. The MONET trial: darunavir/ritonavir with or without nucleoside analogues, for patients with HIV RNA below 50 copies/ml. AIDS. 2010 Jan 16;24(2):223-30. doi: 10.1097/QAD.0b013e3283348944. PMID 20010070
- [Background] Mathis S, Khanlari B, Pulido F, Schechter M, Negredo E, Nelson M, Vernazza P, Cahn P, Meynard JL, Arribas J, Bucher HC. Effectiveness of protease inhibitor monotherapy versus combination antiretroviral maintenance therapy: a meta-analysis. PLoS One. 2011;6(7):e22003. doi: 10.1371/journal.pone.0022003. Epub 2011 Jul 19. PMID 21811554
- [Background] Gilks CF, Walker AS, Dunn DT, Gibb DM, Kikaire B, Reid A, Musana H, Mambule I, Kasirye R, Robertson V, Ssali F, Spyer M, Pillay D, Yirrell D, Kaleebu P; DART Virology Group and Trial Team. Lopinavir/ritonavir monotherapy after 24 weeks of second-line antiretroviral therapy in Africa: a randomized controlled trial (SARA). Antivir Ther. 2012;17(7):1363-73. doi: 10.3851/IMP2253. Epub 2012 Jul 19. PMID 22814125
- [Background] Bartlett JA, Ribaudo HJ, Wallis CL, Aga E, Katzenstein DA, Stevens WS, Norton MR, Klingman KL, Hosseinipour MC, Crump JA, Supparatpinyo K, Badal-Faesen S, Kallungal BA, Kumarasamy N. Lopinavir/ritonavir monotherapy after virologic failure of first-line antiretroviral therapy in resource-limited settings. AIDS. 2012 Jul 17;26(11):1345-54. doi: 10.1097/QAD.0b013e328353b066. PMID 22441252
- [Background] Castagna A, Danise A, Menzo S, Galli L, Gianotti N, Carini E, Boeri E, Galli A, Cernuschi M, Hasson H, Clementi M, Lazzarin A. Lamivudine monotherapy in HIV-1-infected patients harbouring a lamivudine-resistant virus: a randomized pilot study (E-184V study). AIDS. 2006 Apr 4;20(6):795-803. doi: 10.1097/01.aids.0000218542.08845.b2. PMID 16549962
- [Background] Bunupuradah T, Chetchotisakd P, Ananworanich J, Munsakul W, Jirajariyavej S, Kantipong P, Prasithsirikul W, Sungkanuparph S, Bowonwatanuwong C, Klinbuayaem V, Kerr SJ, Sophonphan J, Bhakeecheep S, Hirschel B, Ruxrungtham K; HIV STAR Study Group. A randomized comparison of second-line lopinavir/ritonavir monotherapy versus tenofovir/lamivudine/lopinavir/ritonavir in patients failing NNRTI regimens: the HIV STAR study. Antivir Ther. 2012;17(7):1351-61. doi: 10.3851/IMP2443. Epub 2012 Jul 2. PMID 23075703
- [Derived] Ciaffi L, Koulla-Shiro S, Sawadogo AB, Ndour CT, Eymard-Duvernay S, Mbouyap PR, Ayangma L, Zoungrana J, Gueye NFN, Diallo M, Izard S, Bado G, Kane CT, Aghokeng AF, Peeters M, Girard PM, Le Moing V, Reynes J, Delaporte E; MOBIDIP study group. Boosted protease inhibitor monotherapy versus boosted protease inhibitor plus lamivudine dual therapy as second-line maintenance treatment for HIV-1-infected patients in sub-Saharan Africa (ANRS12 286/MOBIDIP): a multicentre, randomised, parallel, open-label, superiority trial. Lancet HIV. 2017 Sep;4(9):e384-e392. doi: 10.1016/S2352-3018(17)30069-3. Epub 2017 May 28. PMID 28566227
- See also: Sponsor site — http://anrs.fr/